CLINICAL TRIAL: NCT01688232
Title: Colorectal Cancer: a Prospective Multicentric Study of the in Situ Immune Infiltrate for the Identification of the Patients at High Risk of Relapse
Brief Title: The Immunoscore as a Prognostic Marker for Patients With a Colorectal Cancer
Acronym: IMMUCOL
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: NI11033
Record Dates: First submitted 2012-09-14; First posted 2012-09-19 (Estimated); Last update posted 2021-10-12 (Actual); Status verified 2021-10

CONDITIONS: Colorectal Cancer; Surgical Resection of the Colorectal Tumor
Keywords: colorectal cancer; tumor resection; immunoscore; lymphocytic density; CD3; CD8; CD45RO; biopsy; genetic feature of the tumor; relapse; immunohistochemistry; image analysis software
MeSH Terms: conditions — Colorectal Neoplasms; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The pathologist of each center will choose a tumor block containing the core of the tumor and the invasive margin. Three tissue sections of 4 microns of this tumor block will be cut and deposited on glass slides for the immunohistochemical analyses. Four tissue sections of 4 microns will be cut and deposited in a safe lock eppendorf tube for a DNA extraction. If biopsies for diagnostic purpose are available in the laboratory of pathology for the same patient, one tissue section of 4 microns of each biopsy will be cut and deposited on a glass slide
Oversight: Data Monitoring Committee: No

SUMMARY:
Medical and Scientific Background: Colorectal cancers (CRC) are the leading cancers in both genders. This cancer is of prognostic severity. The prognosis of this cancer has not been significantly improved. The treatment of colonic cancer is primarily based on surgery. Adjuvant chemotherapy is proposed for metastatic cancers (stages III and IV). However nearly 30% of patients with localized cancer (stage II) will present a recurrence. Despite intense research efforts, no markers of sufficient prognostic value (independent of TNM) are available to identify this group of patients and justify intensified therapy. The natural history of cancer involves interactions between the tumor and the immune system of the host. The immune infiltration at the tumor site may be indicative of host response. We showed that the density of intratumor memory T cells (CD45RO) and cytotoxic T cells (CD8) in tumor regions (the core and the invasive margin) influenced the occurrence of early events of metastasis (tumor emboli) and was strongly associated with prognosis of patients with CRC (Pagès et al, NEJM-2005). This immune criterion was a better predictor of survival than the "gold standard" histoprognostic data of tumor invasion (T stage and N) and allowed to identify a group of patients at high risk of recurrence (*2). The availability of this immune criterion in clinical practice could improve the prognostic assessment of patients and better guide the therapeutic. A dedicated platform has been implemented in our hospital to speed up the transfer of this immune investigation into the clinic. The investigation takes into account the density of immune cell populations in tumor regions (the core and the invasive front of the tumor). This methodology has been validated for the markers CD45RO, CD3 and CD8 and leads to the creation of an immune score ("immunoscore" ranging from IO to I4). We validated the prognostic impact of the immunoscore in a retrospective series of 250 colorectal cancers. The main objective of this multicentric prospective clinical study is to assess in clinical practice the "immunoscore" and measure its prognostic value. The cohort study will include 400 patients with CRC stage I to IV (6 centers for inclusion; Paris-HEGP, Dijon, Bobigny-Avicenne, Besancon, Poitiers, Rouen). Two years of inclusion and a follow-up of 3 years for each patient will be performed (co-financing for data collection during the 4th and 5th year planned). For each patient, the pathologist of the center will send to the immunomonitoring platform of HEGP tissue sections from a paraffin block containing the tumor regions. The investigations will combine a step of immunostaining for CD3, CD8, and CD45RO (Ventana automate) markers, high-resolution scanning of the stained slides and quantification of digital images by an imaging module developed by our group from the program of Developer XD of Définiens company. The immunoscore will be calculated and the score will be correlated to the clinical data for the relapse and the survival. The secondary objective of this program is to evaluate the prognostic performance of the immune infiltrate on the biopsies performed for diagnostic purposes. This study will be conducted on patients of the cohort whose biopsies were performed in the same hospital than surgery and whose samples are available in pathology laboratories involved (representing 50% of cases). For the same patients will be conducted a genetic investigation of the tumor to assess the MSI status, the presence of a K-Ras and BRAF mutations. This investigation will be performed on tumor sections from the same tumor block selected for the immunohistochemical analyses. The sections will be processed by the Department of Biology, Hôpital Européen Georges Pompidou. The prognostic performance of the immune investigations performed on tumor sections and biopsies will be compared to that of genetic features of the tumor. Finally, a questionnaire will be sent every six months along the monitoring of the patients to obtain information concerning (i) the emergence of an immune disorder (such as allergy, autoimmunity, inflammatory process) and (ii) the psychological status of the patients. The potential impact of such parameters during the course of the disease on the prediction of the relapse and survival obtained with the immunoscore performed at the time of surgery will be evaluated. Expected results : This prospective study is an indispensable step for the clinical validation of the prognostic value of the immunoscore. The secondary objectives should help to precise the benefit of a concomitant analysis of the biopsy, the genetic features of the tumor. The questionnaire should help to identify the clinical parameters to track along the monitoring

DETAILED DESCRIPTION:
The main objective is to assess the impact of the immunoscore in the clinical practice. To this end, the immune parameter (CD3, CD8, CD45RO) of colorectal cancers (stage I-IV) will be evaluated prospectively through a large multicenter study. 400 patients with CRC stage I to IV will be included (6 centers for inclusion; Paris-HEGP, Dijon, Bobigny-Avicenne, Besancon, Poitiers, Rouen). The number of patients to be included has been calculated on the basis of an inclusion period of 24 months, a follow-up of 3 years (a collection of data during the 4th and 5th year is planned with a co-financing), an expected event rate of 20%, a prognostic value of the immune parameter similar to that observed in the retrospective study of 399 patients with CRC (*1) and a power of the test of 90%. During both initial management and follow-up, all therapeutic procedures will be registered (surgery, radiotherapy, chemotherapy…). Data will be collected from clinical examination, radiological exams and biological tests that are usually performed during a hospitalization for colorectal cancer: Full clinical examination and questioning about the presence of personal and family history of CRC, adenomas and other cancers; Abdominal ultrasound, chest X-ray; Computed tomography (CT) and magnetic resonance imaging (MRI) according to clinician's requirement; Standard laboratory tests and blood assay for carcinoembryonic antigen (CEA); The Histopathologic study of the tumor containing the status of the surgical excision margins, the histological type of cancer, the level of parietal invasion, the number of lymph nodes examined and the number of metastatic lymph nodes, according to the TNM classification. Patients will be followed-up every 3 months during the first 2 years, and every 6 months for the rest of the follow-up period, as recommended. Each patient will be followed up to 5 years. Clinical, biological and radiological data will be registered into a specific CRF. Verification of inclusions and monitoring of data will be conducted by the HEGP Clinical Research Unit (URC HEGP) and the principal investigator. A plan for data-management will be built in line with the monitoring. A questionnaire will also be sent to the patients every six month for five years. This questionnaire was built by Pr F Pagès and by psychologists and psychiatrists to search for information concerning (i) the presence of an immune disorder (such as allergy, autoimmunity, inflammatory process) and (ii) the psychological status of the patients (eg. depression). After monitoring, all data will be stored using a double data entry system in a MS-Access database designed by the URC-HEGP and in the TME.dB database created by the team of the principal investigator. The 2 databases will be merged, and the final data base will be frozen for statistical analysis. Sample preparation: The pathologist of each center will choose a tumor block containing the core of the tumor and the invasive margin. This tumor block is part of the tumor samples routinely processed by the department of Pathology for diagnosis. three tissue sections of 4-microns will be made and deposit on a glass slide to perform the immunohistochemistry. Four tissue sections of 4-microns will be made and deposit on an Eppendorf safe lock tubes to perform the genetic analyses. Anonymous patient names on the slides and tubes will be provided by using a code number and initials of the patient. If biopsies for diagnostic purposes are available (i.e. those performed for the patients during their initial hospitalization (50% of cases), A tissue sections of each biopsy will be done. All slides and tubes will be sent by mail to the HEGP platform for analysis of the immune infiltrate and to the Biology department for the genetic analyses. The immunoscore will be determine using the following steps: Immunostainings for CD3, CD8, CD45RO on Benchmark XT automate; Scanning the immunostainings on Hamamatsu scanner: Quantification of the immune populations in specific tumor areas (the core and the invasive margin) with a dedicated image analysis module based on the recognition of histological structures adapted to colorectal cancer. This module has been developed by our group in connection with the Definiens company. A semi-automatic procedure allows the quantification of stained cells in each tumor region. Each region is divided into tiles of 800 microns side (500 to 700 tiles analyzed per tumor). The density of each marker is calculated using the mean density of the three tiles the most infiltrated in each tumor region. A categorization into high density (Hi) or low (Lo) for each marker in each tumor region of interest will be performed. This categorization is done by comparing the observed density with the optimal cut-off density (min p value approach) we previously determined for the DFS and OS in a retrospective study of 250 CRC. Genetic analyses: The tubes containing the sections for the genetic analyses of patients with inform consent signed for genetic investigation will be transfer to the Department of Biology, Hôpital Européen Georges Pompidou. The % of tumor cells of each specimen will be determined by a pathologist (based on a H&E evaluation; less than 10%, 10-20%, 20-50%, up to 50% tumor cells) and the DNA extraction will be performed. Genetic investigation will comprise the MSI status, the presence of a K-Ras and BRAF mutation

ELIGIBILITY:
Inclusion Criteria:

* Adult patient with newly diagnosed colorectal cancer.
* Patient with signed informed consent.
* Follow up made by the clinical center for inclusion or by a medical team in relation with the center.

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patient with newly diagnosed colorectal cancer.
Sampling Method: Non-Probability Sample
Enrollment: 459 (Actual)
Dates: Start 2012-09-27 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
relapse in relation with the immunoscore determined on a tumor section. | evry 3 month during 3 years and every six months during the fourth year
  this primary outcome (relapse) will be correlated to the immunoscore determined in the primary tumor (eg. the density of immune cells in tumor regions)

SECONDARY OUTCOMES:
relapse in relation with the immunoscore on biopsies | evry 3 month during 3 years and every six months during the fourth year
  this primary outcome (relapse) will be correlated to the immunoscore determined in biopsies performed for diagnosis purpose (eg. the density of immune cells in the biopsies specimens)
relapse in relation with the genetic features of the tumor | evry 3 month during 3 years and every six months during the fourth year
  this primary outcome (relapse) will be correlated to the genetic features of the tumor (eg. MSI status, K-Ras and BRAF mutations). The prognostic performance of the genetic and immunologic analyses will be compared.
relapse in relation with the immunological events and psychological status of the patient during the monitoring | every six months during 4 years
  a questionnaire will be sent every six months along the monitoring of the patients to obtain informations concerning (i) the emergence of an immune disorder and (ii) the psychological status of the patients. The potential impact of such parameters during the course of the disease on the prediction of the relapse and survival obtained with the immunoscore performed at the time of surgery will be evaluated. The questionnaire should help to identify the clinical parameters to track along the monitoring.

CONTACTS AND LOCATIONS:
Overall Officials: Franck Pagès, Professor (MD-PHD), Principal Investigator — AP-HP; Paris Descartes University
Locations (6):
- France (6):
  - Hopital de Besançon (CHU), Besançon
  - Hopital Avicenne (CHU), Bobigny
  - Hopital de Dijon (CHU), Dijon
  - Hopital Europeen Georges Pompidou (HEGP), Paris
  - Hopital de Poitiers (CHU), Poitiers
  - Hopital Charles Nicolle(CHU), Rouen

REFERENCES:
- [Result] Galon J, Costes A, Sanchez-Cabo F, Kirilovsky A, Mlecnik B, Lagorce-Pages C, Tosolini M, Camus M, Berger A, Wind P, Zinzindohoue F, Bruneval P, Cugnenc PH, Trajanoski Z, Fridman WH, Pages F. Type, density, and location of immune cells within human colorectal tumors predict clinical outcome. Science. 2006 Sep 29;313(5795):1960-4. doi: 10.1126/science.1129139. PMID 17008531
- [Result] Pages F, Kirilovsky A, Mlecnik B, Asslaber M, Tosolini M, Bindea G, Lagorce C, Wind P, Marliot F, Bruneval P, Zatloukal K, Trajanoski Z, Berger A, Fridman WH, Galon J. In situ cytotoxic and memory T cells predict outcome in patients with early-stage colorectal cancer. J Clin Oncol. 2009 Dec 10;27(35):5944-51. doi: 10.1200/JCO.2008.19.6147. Epub 2009 Oct 26. PMID 19858404
- [Result] Mlecnik B, Tosolini M, Kirilovsky A, Berger A, Bindea G, Meatchi T, Bruneval P, Trajanoski Z, Fridman WH, Pages F, Galon J. Histopathologic-based prognostic factors of colorectal cancers are associated with the state of the local immune reaction. J Clin Oncol. 2011 Feb 20;29(6):610-8. doi: 10.1200/JCO.2010.30.5425. Epub 2011 Jan 18. PMID 21245428